CLINICAL TRIAL: NCT05065229
Title: A Study of Agreement Between Oxygen Saturation Measured by Two Probes in Infants on the Neonatal Unit
Acronym: Ag-OS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: IRAS 297715
Record Dates: First submitted 2021-08-04; First posted 2021-10-04 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Neonatal Disease
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Intervention Model Description: Parallel group, randomised study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A computer-generated random number sequence will be obtained to determine which probe is attached to which foot. The sequence will be kept in opaque, sequentially numbered envelopes that will be opened just before the probes are attached to the feet of the participant. The clinical team nurse who will record the oxygen saturation readings will be blinded to which probe is attached to which foot by covering the feet securely after the probes have been attached. The probes will be designated as A and B. The study statistician will be blind to which probe is A and which is B until all data analyses are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Right foot no.520 Left foot no.521
  Interventions: Device: Oxygen saturation probe Mindray 520 N and Mindray 521 N
- B (Experimental): Right foot no.521 Left foot no.520
  Interventions: Device: Oxygen saturation probe Mindray 520 N and Mindray 521 N

INTERVENTIONS:
Device: Oxygen saturation probe Mindray 520 N and Mindray 521 N — Two oxygen saturation probes will be used in this study:
  Mindray 520 N is a disposable oxygen saturation sensor for neonates and adults. It is a disposable, single-use sensor that is wrapped around the infant's arm or foot. Its ends stick together giving a firm, close contact with the skin.
  Mindray 521 N is another disposable oxygen saturation sensor for neonates and adults that is used on the neonatal unit in routine practice. As Mindray 520 N and 521 N are CE marked and used within their intended purposes we do not require a letter of no objection from the MHRA for that usage. The Mindray probes will be used without modification and there are no safety issues to the patient. Therefore, a letter of no objection from the MHRA is not required and this is not a medical device study under the Medical Devices Directive.

SUMMARY:
On the neonatal unit in Derby, two types of probes are in routine use: Mindray 520 N and Mindray 521 N. Feedback from parents and staff show that there are concerns that the two probes given very different oxygen saturation readings and, often, do not agree with each other. This has raised concerns that infants' clinical care may be affected by the choice of probe. It is important to know if the two probes give similar results or not to ensure that infants get the appropriate monitoring and respiratory support as needed for good neonatal care. In this study, we will compare the reading made by the two probes and determine whether the readings of the two probes agree with each other and if any disagreement is such that clinical decision making is affected by the difference.

DETAILED DESCRIPTION:
Continuous monitoring of oxygen saturation level is a key component of neonatal intensive care and NICE recommends that all neonatal services "ensure that systems are in place for preterm babies to have a target saturation level of 91% to 95%" and that this is monitored using "continuous pulse oximetry" (NICE Quality statement 4 in Quality Standard QS193: https://www.nice.org.uk/guidance/qs193/chapter/Quality-statement-4-Oxygen-saturation). Oxygen saturation monitoring is used to provide optimal respiratory support to preterm infants to ensure adequate oxygenation of tissues while preventing risks of conditions such as retinopathy of prematurity and bronchopulmonary dysplasia [1]. It is equally important in term born infants who require intensive care such as for determining adequate oxygenation for respiratory support and screening for congenital heart disease [2]. For these reasons, most infants in neonatal units are continuously monitored using pulse oximetry, a simple and painless test that measures blood oxygen levels by passing a small beam of light through the infant's hand or foot. This measures the changes in light absorption to calculate the levels of oxygenated and deoxygenated blood. To do this the light (or probe) has to be attached to the infant's hand or foot using a tie or a sticker. The probe must be attached firmly for the saturation monitor to pick up the correct readings. As neonatal skin is delicate and it is often difficult to stick objects to it, neonatal oxygen saturation probes are carefully designed. Many different types of saturation probes are in routine use in neonatal units. It is important to ensure that they give accurate and comparable readings. In the neonatal unit in Derby, two types of probes are in routine use: Mindray 520 N and Mindray 521 N. Feedback from parents and staff show that there are concerns that the two probes given very different oxygen saturation readings and, often, do not agree with each other. This has raised concerns that infants' clinical care may be affected by the choice of probe. It is important to know if the two probes give similar results or not to ensure that infants get the appropriate monitoring and respiratory support as needed for good neonatal care. In this study, we will compare the reading made by the two probes and determine whether the readings of the two probes agree with each other and if any disagreement is such that clinical decision making is affected by the difference.

ELIGIBILITY:
Inclusion Criteria:

* Infants who need oxygen saturation monitoring for clinical care
* Infants born preterm (<37 weeks' gestation) who are < 7 days of age and need respiratory support including supplemental oxygen
* Infants born preterm (<37 weeks' gestation) who are in supplemental oxygen at >34 weeks' gestation
* Infants born at term gestation (< 37 weeks' gestation) who require respiratory support including supplemental oxygen
* Infants with suspected cardiac disease

Exclusion Criteria:

* Infants who have intravenous or arterial lines attached to either foot.
* Infants who have any condition that may cause differential oxygen saturation or blood flow to the lower limbs such as venous thrombosis.
* Infants who have local infections or skin lesions on either foot.
* Infants older than 5 months of age

Ages: 32 Weeks to 60 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-14 (Actual)

PRIMARY OUTCOMES:
oxygen saturation of babies using Minday 520 N and Minday 521 N | 12 months
  Oxygen saturation readings using Minday 520 N and Minday 521 N probes simultaneously

SECONDARY OUTCOMES:
clinical decision making | 12 months
  clinical decisions made, such as giving supplemental oxygen to infants on the neonatal unit following oxygen saturation readings from Minday 520 N and Mindray 521 N

CONTACTS AND LOCATIONS:
Overall Officials: shalini ojha, Principal Investigator — University of Nottingham
Locations (1):
- University Hospitals of Derby and Burton, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No